CLINICAL TRIAL: NCT01000142
Title: Preventative OMT and the Nursing Home Patient
Brief Title: Preventative Osteopathic Manipulative Treatment (OMT) and the Nursing Home Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 501-332
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: General Health Status
Keywords: Osteopathic; Manipulation; Preventative; Elderly; Nursing Home; Prevention: General Health Status
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment as Usual Control Group (No Intervention)
- Light Touch Group (Sham Comparator): Focused osteopathic musculoskeletal exam; contact ribs to simulate rib raising and paraspinal muscle inhibition; contact lower rib margin to simulate abdominal diaphragm release; palpate the four quadrants of the abdomen to simulate abdominal mesenteric/colon release; contact shoulders to simulate thoracic inlet release; contact suboccipital region to simulate thoracic inlet release.
  Interventions: Procedure: Light Touch
- Standard OMT Group (Experimental)
  Interventions: Procedure: Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Focused osteopathic musculoskeletal exam; paraspinal muscle inhibition and/or soft tissue kneading or stretching; rib raising and or rib mobilization; abdominal diaphragm release technique; abdominal mesenteric/colon release; thoracic inlet release technique; hip flexion/extension range of motion; shoulder range of motion with pectoral traction; cervical paraspinal muscle inhibition and/or soft tissue kneading or stretching; suboccipital release technique; specific OMT of significant somatic dysfunction (variable).
  Other Names: OMT; OMM; Osteopathic Manipulative Medicine; Manipulation
  Arms: Standard OMT Group
Procedure: Light Touch — Focused osteopathic musculoskeletal exam; contact ribs to simulate rib raising and paraspinal muscle inhibition; contact lower rib margin to simulate abdominal diaphragm release; palpate the four quadrants of the abdomen to simulate abdominal mesenteric/colon release; contact shoulders to simulate thoracic inlet release; contact suboccipital region to simulate thoracic inlet release.
  Other Names: Sham manipulation; Placebo manipulation
  Arms: Light Touch Group

SUMMARY:
This pilot research study will investigate the possible benefit that elderly nursing home patients may receive from regular Osteopathic Manipulative Medicine (OMM) care during the winter months. The study is based on the osteopathic philosophies that structure and function are interrelated and that the body has self-healing mechanisms. The body is expected to have optimized ability to heal itself "when all its parts are in place" (AT Still). This study is looking at subject population for whom their ability to take care of themselves is diminished by their underlying diseases. Based on the osteopathic philosophies, optimization of the nursing home patient's physical structure through osteopathic manipulative treatment (OMT) should enhance their body's homeostatic mechanisms. This study is assessing the validity of these philosophies by looking at the effect of OMT on the global health of these individuals.

DETAILED DESCRIPTION:
This study will randomly assign 36 nursing home patients from two Kirksville nursing homes into three groups of twelve subjects: 1) treatment as usual (TAU) control group; 2) light touch (LT) group, and 3) standard OMT group.

This study will begin with rolling admission of volunteer nursing home patients starting in October 2009. Subjects in the LT and OMT group would receive focused musculoskeletal evaluations twice a month for 5 months (10 visits). The OMT group would also receive an OMT protocol each visit that would specifically address optimization of homeostatic mechanisms - balancing autonomic nervous system and improving lymphatic drainage- along with OMT that would specifically target somatic dysfunction found on that day's evaluation. The LT group subjects would receive a light touch protocol meant to simulate OMT. The TAU group will receive no intervention. The protocol period will end for all subjects by March 2010. All osteopathic examinations, assessments, and treatments will be performed at the participating nursing homes.

Throughout the protocol period, at the end of the winter (March 2010), and three months later (June 2010), retrospective chart reviews will be conducted on all subjects. All cause morbidity and mortality for all subjects will be assessed by monitoring their medications, health history changes, and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Participating Nursing Home
* Life Expectancy of at Least 6 Months

Exclusion Criteria:

* Diagnosis of Terminal Cancer
* Diagnosis of Active Tuberculosis
* Diagnosis of Metabolic Bone Disease or Condition That Would Place Patient at Risk for Pathological Fracture
* Unable to Cooperate
* Unable to Tolerate OMT
* OMT is Contraindicated

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in subject health status: reviewing data regarding medication usage, co-morbidities, hospitalizations and activities of daily living. | Five Months

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Snider, DO, Principal Investigator — A.T. Still University-Kirksville College of Osteopathic Medicine
Locations (2):
- United States (2):
  - Kirksville Manor Care Center, Kirksville, Missouri
  - Twin Pines Adult Care Center, Kirksville, Missouri

REFERENCES:
- [Derived] Snider KT, Snider EJ, Johnson JC, Hagan C, Schoenwald C. Preventative osteopathic manipulative treatment and the elderly nursing home resident: a pilot study. J Am Osteopath Assoc. 2012 Aug;112(8):489-501. PMID 22904246